CLINICAL TRIAL: NCT04850625
Title: Pyrotinib Plus Vinorelbine Versus Lapatinib Plus Capecitabine in Patients With Previously Treated HER2-Positive Metastatic Breast Cancer: a Multicenter, Retrospective Study
Brief Title: Pyrotinib Plus Vinorelbine Versus Lapatinib Plus Capecitabine
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-14
Record Dates: First submitted 2021-04-16; First posted 2021-04-20 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: Pyrotinib; Lapatinib; Vinorelbine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pyrotinib Plus Vinorelbine: lapatinib (750-1,250 mg/day) plus capecitabine (1,500-2,000 mg/m2)
- Lapatinib Plus Capecitabine: pyrotinib (320-400 mg/day) plus vinorelbine (25mg/ m2 intravenously or 60 mg/m2 orally on days 1 and 8 per 21 days)

SUMMARY:
Pyrotinib Plus Vinorelbine Versus Lapatinib Plus Capecitabine

DETAILED DESCRIPTION:
This is a retrospective study aiming to explore the efficacy and safety of Pyrotinib plus Vinorelbine versus Lapatinib plus Capecitabine in patients with previously treated HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* HER2+ MBC patients scored +3 by immunohistochemical (IHC) analysis or scored +2 and the result of fluorescence in situ hybridization was positive.
* Patients were previously treated with trastuzumab in the advanced setting and a taxane in any setting.
* Patients received lapatinib (750-1,250 mg/day) plus capecitabine (1,500-2,000 mg/m2) or pyrotinib (320-400 mg/day) plus vinorelbine (25mg/ m2 intravenously or 60 mg/m2 orally on days 1 and 8 per 21 days) for at least one cycle, starting from Jun 2015 to Jan 2021.
* Patients had complete medical records. All data were retrospectively collected from medical records of individual institutions.

Exclusion Criteria:

* Incomplete medical history

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided